CLINICAL TRIAL: NCT03366896
Title: Validation Study of the Malay Version of the 3-Minute Diagnostic Interview for Confusion Assessment Method Defined Delirium (3D-CAM)
Brief Title: Validation Study of the Malay Version of 3D-CAM
Acronym: VS-MEDCAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Chin Yi Zhe, Dr, University of Malaya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MEDCAM1
Record Dates: First submitted 2017-12-03; First posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Postoperative Delirium; Diagnosis, Psychiatric
MeSH Terms: conditions — Emergence Delirium; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Delirium (Experimental): Diagnosis of delirium according to 5th Edition of The Diagnostic and Statistical Manual of Mental Disorders (DSM-5) by Psychiatrist.
  Interventions: Diagnostic Test: Malay 3D-CAM diagnostic tool 1; Diagnostic Test: Malay 3D-CAM Diagnostic tool 2

INTERVENTIONS:
Diagnostic Test: Malay 3D-CAM diagnostic tool 1 — Assessor 1 uses Malay 3D-CAM to detect Delirium
Diagnostic Test: Malay 3D-CAM Diagnostic tool 2 — Assessor 2 uses Malay 3D-CAM to detect Delirium

SUMMARY:
Validation of the Malay version of 3D-CAM, involving two-staged process.

1. Translation and cultural adaptation of 3D-CAM into the Malay language.
2. Testing for Validity and Reliability of the translated 3D-CAM tool to detect postoperative delirium.

DETAILED DESCRIPTION:
1. Translation and Cultural Adaptation

   The research panel, who consisted of experts in the clinical field of anesthesia, did the meticulous process of translation and cultural adaptation of 3D-CAM.

   This process included independent translation by the research panel, reconciliation of two independent translated 3D-CAM, ethics approval prior to pilot study on 20 relevant subjects, back translation into English and finalizing the Malay version of 3D-CAM for the next phase of testing.
2. Testing for Validity and Reliability of the translated 3D-CAM tool

Patients were recruited pre-operatively after reading the patient's information sheet and signing the informed consent.

Post-operatively, two trained assessors separately administered the Malay 3D-CAM on the recruited patients. One of the trained assessors administered the original 3D-CAM on the same patients at a different time. Standard reference of diagnosing delirium was made by a psychiatrist using the DSM V criteria, after interviewing the patients.

1. For validity, the diagnosis of delirium made using the Malay 3D-CAM tool was tested against the standard reference for diagnosing delirium according to the DSM V criteria made by a psychiatrist
2. For inter-rater reliability, the diagnosis of delirium made by two trained assessors using the Malay 3D-CAM tool were statistically compared.
3. For parallel reliability, the diagnosis of delirium made using the Malay 3D-CAM was compared to the original English version of 3D-CAM.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years old and above
* Patients undergoing non-cardiac surgery

Exclusion Criteria:

* Patients undergoing cardiac Surgery
* Unable to communicate in the Malay Language
* Patients who were in the intensive care unit peri-operatively
* Patients whose surgery was cancelled
* Patients who were deaf and dumb
* Patients who had been diagnosed as delirious or has psychosis history before assessment
* Glasgow Coma Scale of < 12 / 15
* Patients who remained comatose throughout the investigation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-06-26 (Actual); Primary Completion 2016-09-26 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Construct Validity | 3 months
  Assess validity of the translated Malay 3D-CAM to Standard Reference for Diagnosis of Delirium

SECONDARY OUTCOMES:
Inter-rater Reliability | 3 months
  Assess the inter-rater reliability of 2 trained assessor using the Malay 3D-CAM
Parallel Reliability | 3 months
  Assess the parallel reliability of using Malay 3D-CAM to the original version of 3D-CAM
Factors associated with post-operative delirium | 3 months
  Assess factors associated with post-operative delirium

CONTACTS AND LOCATIONS:
Overall Officials: Chew Yin Wang, MBChB, FRCA, Study Chair — Professor University Malaya Anaesthesiology Department; Pui San Loh, MBBS, FANZCA, Principal Investigator — Consultant University Malaya Anaesthesiology Department; Yi Zhe Chin, MB BCh, MCAI, Principal Investigator — Master Student University Malaya Anaesthesiology Department; Chong Guan Ng, MPM,MSc,PhD, Principal Investigator — Associate Professor University Malaya Consultant Psychiatrist

IPD SHARING:
Plan to Share IPD: Undecided
Individual responses from the Malay 3D-CAM